CLINICAL TRIAL: NCT03038724
Title: Randomised Study Comparing Two HIV Screening Strategies in the Emergency Department Using an Electronic Tablet Questionnaire: The PETTSEQ Study (PErformance of Two Testing Strategies by Electronic Questionnaire)
Brief Title: Randomised Study Comparing Two HIV Screening Strategies
Acronym: PETTSEQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Olivier Hugli, Head Physician, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CHUV
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infections
Keywords: HIV testing
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Randomised, single-blind study
Who Masked: Care Provider, Investigator
Masking Description: The study investigator will not know which arm each patient is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted testing (Other): Patients complete a questionnaire on risk factors for HIV acquisition and are offered rapid (fingerprick) HIV testing if their questionnaire responses indicate they have HIV risk factors
  Interventions: Diagnostic Test: Rapid HIV test
- Non-targeted screening (Other): Patients offered a brief information on HIV and HIV testing and are then offered rapid (fingerprick) HIV testing without completing an HIV risk factor assessment
  Interventions: Diagnostic Test: Rapid HIV test

INTERVENTIONS:
Diagnostic Test: Rapid HIV test
  Other Names: INSTI

SUMMARY:
A randomised, single-blind study (the study investigator will not know which arm each patient is assigned to) conducted to examine the most effective strategy for conducting HIV testing in the Emergency Department (ED) using an electronic tablet. The study will take place in the ED at Lausanne University Hospital (LUH) between August and December 2015 in the context of the Masters project of a medical student studying at the Faculty of Medicine at Lausanne University.

DETAILED DESCRIPTION:
In Switzerland, the national HIV testing recommendations have proposed targeted and diagnostic HIV testing since 2007. These recommendations list medical conditions and populations at risk in which HIV testing is indicated. The difficulty with this targeted approach is that it relies on medical personnel 1) to be aware that the medical conditions listed have an association with HIV infection and 2) to be able to identify their patients as coming from at-risk populations. In other countries, notably the United States, France and the United Kingdom, national HIV testing recommendations propose non-targeted screening whereby everyone presenting to a medical facility is tested if the HIV seroprevalence in the catchment population is above a defined threshold (0.1% for the US and France; 0.2% for the UK). As HIV seroprevalence in Switzerland already exceeds these thresholds, the current study will be performed to see whether non-targeted HIV testing using electronic tablets is acceptable and feasible in our Emergency Department (ED).

ED patients will be randomised to a targeted or non-targeted arm after consenting to participate. Eighty patients will be assigned to each study arm. Participating patients will be issued with an electronic tablet and invited to follow the instructions on the screen. Targeted arm patients will be invited to complete a questionnaire on HIV risk factors and, if one or more risk factors are present, they will be informed that HIV testing is indicated and will be invited to take a free rapid HIV test. Non-targeted arm patients will be provided with information about HIV and HIV testing and will then be invited to take a free rapid HIV test without any questions regarding risk factors. Patients in each arm who are either not offered (targeted arm) or who decline rapid testing (non-targeted arm) will undergo secondary cross-screening in which targeted arm patients will be automatically directed by the tablet to the non-targeted arm information page and non-targeted arm patients will be directed to the targeted arm questionnaire. The primary endpoint is patient acceptance of HIV testing. The secondary objective is to examine the effect of cross-screening strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 and ≤ 75 years old
* Patients admitted to an ED examination cubicle within the preceding 12 hours

Exclusion Criteria:

* Patients clinically unstable (admitted to resus or considered unstable by the treating ED doctor)
* Patients transferred from another hospital
* Patients unable to provide informed consent (for example, through cognitive impairment, acute alcohol intoxication or intoxication by opiates or other psycho-active substances, acute psychosis, being hard of hearing or not French-speaking and with no interpreter)
* Patients of known HIV+ status
* Patients who have already been offered HIV screening during their ED visit by the treating ED doctor prior to enrolment in the study
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2015-11-28 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Patient acceptance of rapid HIV testing in the ED | 4 months
  Patient acceptance of rapid HIV testing when offered by electronic questionnaire

SECONDARY OUTCOMES:
HIV testing rate after cross-screening strategy | 4 months
  HIV testing accepted when patients without risk factors are offered testing or if patients offered testing without risk factor assessment then complete an assessment which shows they have risk factors for HIV acquisition

OTHER OUTCOMES:
Ease of use of electronic questionnaire | 4 months
  Degree of assistance required by patients when they use the electronic tablet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillet C, Darling KEA, Senn N, Cavassini M, Hugli O. Targeted versus non-targeted HIV testing offered via electronic questionnaire in a Swiss emergency department: A randomized controlled study. PLoS One. 2018 Mar 7;13(3):e0190767. doi: 10.1371/journal.pone.0190767. eCollection 2018. PMID 29513659